CLINICAL TRIAL: NCT03652272
Title: Development and Evaluation of an Electronic Health Record-based Medication Complete Communication (EMC2) Strategy (Phase 2)
Brief Title: Development and Evaluation of an Electronic Health Record-based Medication Complete Communication (EMC2) Strategy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Principal Investigator, Michael S. Wolf, Associate Vice Chair for Research, Department of Medicine, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: STU00207507
Record Dates: First submitted 2018-08-28; First posted 2018-08-29 (Actual); Results first posted 2025-03-07 (Actual); Last update posted 2025-03-07 (Actual); Status verified 2025-02

CONDITIONS: Medication Adherence
Keywords: medication safety; adherence; electronic health record
MeSH Terms: conditions — Medication Adherence

STUDY DESIGN:
Intervention Model Description: 2-arm, multi-site, physician-randomized pragmatic trial to evaluate the impact and scalability of the Phase I EMC2 strategy to promote safe medication use and adherence.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EMC2 (Experimental): Following patient movement through a provider visit, the following activities will occur for a select list of pre-specified medications:
  1. Prescribers will receive a 'Best Practices Alert' which recommends patient counseling on medication use and provides an overview of key medication risks
  2. Patients will receive a Medication Guide + Summary with their After Visit Summary
  3. Patients will be asked to complete a brief questionnaire on medication use via the patient portal post visit (at both 1 week and 1 month post visit for this phase of the study)
  4. Portal assessment results and feedback will be provided to the clinic via an inbox message. Clinic staff will respond to any identified problems according to their own clinical care protocols.
  Interventions: Behavioral: EMC2
- Usual Care (No Intervention): Usual care includes 1) variable provider counseling with limited or variable EHR notifications or counseling support; 2) no distribution of print medication information materials, including FDA Medication Guides in clinics and variable distribution in pharmacies; and 3) limited or no active surveillance of medication use post-visits.

INTERVENTIONS:
Behavioral: EMC2 — 1. Prescribers will receive a 'Best Practices Alert' which recommends patient counseling on medication use and provides an overview of key medication risks
  2. Patients will receive a Medication Guide + Summary with their After Visit Summary
  3. Patients will be asked to complete a brief questionnaire on medication use via the patient portal post visit (at both 1 week and 1 month post visit for this phase of the study)
  4. Portal assessment results and feedback will be provided to the clinic via an inbox message. Clinic staff will respond to any identified problems according to their own clinical care protocols.
  Arms: EMC2

SUMMARY:
There is a well-documented need for effective interventions that can help patients understand and safely adhere to prescribed medications, particularly those with greater potential for harm if not taken correctly. The investigators will leverage health and consumer technologies with their EHR-based Medication Complete Communication (EMC2) Strategy to: 1) inform patients about medication risks and safe use, 2) promote provider education and counseling about prescribed drugs and 3) monitor patient adherence outside of visits. The EMC2 Strategy could be feasible, sustainable, and readily available to ambulatory care practices.

DETAILED DESCRIPTION:
This is a 2-arm, multi-site, physician-randomized pragmatic trial to evaluate the impact and scalability of the EMC2 strategy to promote safe medication use and adherence.

Treatment Arms and Duration:

Usual Care. Usual care includes 1) variable provider counseling with limited or variable EHR notifications or counseling support; 2) no distribution of print medication information materials, including FDA Medication Guides in clinics and variable distribution in pharmacies; and 3) limited or no active surveillance of medication use post-visits.

Intervention: EMC2 Strategy.

In brief, there are several components to this strategy that will be embedded into the workflow via EHR/patient portal platforms, mostly automating their implementation. Following patient movement through a provider visit, the following activities will occur for a select list of pre-specified medications:

1. Physician Medication Alert: If a prescribing physician attempts to place a new order or change to an existing study medication prescription, an EHR-generated alert will notify the provider that the medication requires patient counseling. Physicians can opt to ignore this alert.
2. Provider Counseling Support: Content from the 1-page, Med Guide Summary will appear on the screen, if selected by the provider, to orient and inform provider-patient discussion.
3. Automated Delivery of Med Guide + Summary: When patients leave an encounter, the medication order in Epic will automatically cue printing of both the 1-page, health literate Med Guide Summary for study medications and a full Med Guide, if applicable (latter is required by FDA for certain medications only, the former designed to enhance comprehension).
4. Follow-Up Portal Questionnaire: Within 1 week post-visit, patients will receive an automated email prompting them to log on to the patient portal. Patients' will be asked to fill out a short set of questions related to medication adherence, and other medication-related concerns (i.e. cost, side effects). If patients have not completed the questionnaire within 2 days, another email reminder will be sent. The information submitted back by the patient will be stored in the EHR. A second questionnaire will be sent 1 month later.

   The addition of the patient portal will provide opportunities to have ongoing communications with their clinic, access to regimen-specific medication information, and to provide a feedback loop informing healthcare providers of safety and adherence-related behaviors and concerns.
5. EHR Inbox Message to Clinic: The results of the patient portal questionnaire will be sent back to the EHR, populating an inbox message notifying the nurse/clinic staff and/or physician if a patient has a medication risk alert, detailing the nature of the issue (i.e. education needed, adherence problem, side effect concerns, etc.). The system will be flexible and allow the clinic to specify actions to be taken according to their workflow preferences; the default plan is that patient contact will be undertaken by nurses/clinic staff involved with care management.
6. Clinic Counseling: If a problem/concern is flagged during the review of the portal questionnaire, there will be an expectation for a clinic staff member to respond to the concern by calling the patient. A general orientation to staff at the clinic will provide guidance on how to perform brief counseling based on each specific clinic protocol.

Number of Patients:

While the expected sample size for this pragmatic study is 300, the investigators will recruit 330 patients (n=165 per site, the investigators anticipate 90% retention among the recruited sample by 3 months (n=297). The investigators therefore will over sample to accommodate some attrition.

ELIGIBILITY:
Inclusion Criteria:

* Patient is age 18 and older
* Patient is English speaking
* Patient is primarily responsible for administering their own medication
* Patient must have received a new or changed prescription for a product(s), identified by Eli Lilly and the study team, within 7 days of recruitment
* Patient must have access to the internet
* Patient must have a patient portal account

Exclusion Criteria:

* Severe, uncorrectable vision
* Severe hearing impairments
* Severe cognitive impairment
* No access to the internet or patient portal account

Providers must meet the following eligibility criteria:

• Resident, Attending Physician or Mid-level provider (NP, PA) working in the NMHC Endocrinology clinic or other study sites during study dates.

*Adults unable to consent, individuals under the age of 18, and prisoners will be excluded from this research.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 301 (Actual)
Dates: Start 2019-02-08 (Actual); Primary Completion 2021-09-27 (Actual); Study Completion 2021-09-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael S Wolf, PhD MPH, Principal Investigator — Northwestern University; Stacy C Bailey, PhD MPH, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No
There is currently no plan to share IPD.

RESULTS

PARTICIPANT FLOW:
Groups:
- EMC2: Following patient movement through a provider visit, the following activities will occur for a select list of pre-specified medications:
  1. Prescribers will receive a 'Best Practices Alert' which recommends patient counseling on medication use and provides an overview of key medication risks
  2. Patients will receive a Medication Guide + Summary with their After Visit Summary
  3. Patients will be asked to complete a brief questionnaire on medication use via the patient portal post visit (at both 1 week and 1 month post visit for this phase of the study)
  4. Portal assessment results and feedback will be provided to the clinic via an inbox message. Clinic staff will respond to any identified problems according to their own clinical care protocols.
  EMC2: 1) Prescribers will receive a 'Best Practices Alert' which recommends patient counseling on medication use and provides an overview of key medication risks 2) Patients will receive a Medication Guide + Summary with their After Visit Summary 3) Patients will be asked to complete a brief questionnaire on medication use via the patient portal post visit (at both 1 week and 1 month post visit for this phase of the study) 4) Portal assessment results and feedback will be provided to the clinic via an inbox message. Clinic staff will respond to any identified problems according to their own clinical care protocols.
Period: Baseline
Arm/Group | EMC2 | Usual Care
Started | 143 | 158
Completed | 143 | 158
Not Completed | 0 | 0
Period: 3 Month
Arm/Group | EMC2 | Usual Care
Started | 143 | 158
Completed | 126 | 143
Not Completed | 17 | 15
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Lost to Follow-up | 16 | 14

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | EMC2 | Usual Care | Total
Number analyzed (Participants) | 143 | 158 | 301
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.58 (13.99) | 53.61 (14.88) | 53.12 (14.44)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: 1 particiant with missing sex data
  Participants
    number analyzed (Participants) | 143 | 157 | 300
    Female | 82 | 95 | 177
    Male | 61 | 62 | 123
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: 3 participants (2 EMC2 and 1 Usual Care) with missing race data
  Participants
    number analyzed (Participants) | 141 | 157 | 298
    Hispanic | 20 | 21 | 41
    Non-Hispanic White | 50 | 82 | 132
    Non-Hispanic Black | 60 | 41 | 101
    Non-Hispanic Others/Multiracial | 11 | 13 | 24
Education [Count of Participants; unit: Participants] — Population: 2 participants with missing education data
  Participants
    number analyzed (Participants) | 142 | 157 | 299
    Less than High School | 10 | 4 | 14
    High School Graduate | 59 | 59 | 118
    College Graduate | 73 | 94 | 167

OUTCOME MEASURES:

1. Primary Outcome: Medication Specific Knowledge
Description: Patients are asked about their medication's 1) indication, 2) risks or warnings (knowledge of risk/warnings, correct or incorrect per item) and 3) side effects (knowledge of at least two side effects, correct or incorrect per item). Correct answers were graded blindly by 2 reviewers and any discordance was resolved by a third pharmacist. Total scores ranged from 0-100, with a higher value associated with a better outcome, that reflects the percent correct of possible points.
Time Frame: Baseline
Population: This trial was conducted at Northwestern Endocrinology and ACCESS Community Health Network. Due to the Covid-19 pandemic and its impact on recruitment (loss of providers, low patient volume, low prescription volume) at ACCESS performance sites, recruitment was halted in March 2021. The effectiveness of the intervention will be only tested on the Northwestern participants due to statistical power. 2 patients from the intervention group were excluded due to missing outcomes data at follow-up.
Measure: Least Squares Mean (95% Confidence Interval); unit: score (0-100)
Arm/Group | EMC2 | Usual Care
Number analyzed (Participants) | 117 | 147
score (0-100) | 63.82 [59.53 to 68.11] | 62.80 [58.80 to 66.80]

2. Secondary Outcome: Medication Adherence- Ask 12
Description: The ASK-12 survey covers three adherence domains: inconvenience/forgetfulness, treatment beliefs and behavior. Scores range from 12-60, with higher scores translating to greater barriers to adherence.
Time Frame: Baseline-3 Months
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | EMC2 | Usual Care
Number analyzed (Participants) | 117 | 147
units on a scale | 22.33 [21.33 to 23.32] | 21.56 [20.64 to 22.48]

3. Secondary Outcome: Medication Adherence - Proper Use
Description: Patients will be asked the last day they took their medication and how. A patient's proper timing (last day and # of times per day), dosing (number of pills per dose), and spacing between doses (for BID, TID medications only) will be coded as correct or incorrect. Patients will be classified as having properly used their medication if they correctly reported all components.
Time Frame: Baseline- 3 Months
Population: The EMC2 Phase 2 Trial is conducted at Northwestern Endocrinology and ACCESS Community Health Network. Due to the Ccovid-19 pandemic and its impact on recruitment (loss of providers, low patient volume, low prescription volume) at ACCESS performance sites, recruitment was halted in March 2021. The Effectiveness of the intervention will be only tested on the Northwestern participants due to statistical power.
Measure: Least Squares Mean (95% Confidence Interval); unit: Probability of Proper Use (Yes)
Arm/Group | EMC2 | Usual Care
Number analyzed (Participants) | 111 | 146
Probability of Proper Use (Yes) | 0.78 [0.62 to 0.88] | 0.62 [0.45 to 0.76]

ADVERSE EVENTS:
Time Frame: Adverse Event data was collected post 3.5 months from EMC2 intervention.
Description: All participants were asked if they had experienced an adverse event to their prescribed medicine at the 3 month phone interview. If participants endorsed yes and provided details, an AE report was generated.
Arm/Group | EMC2 | Usual Care
All-Cause Mortality (participants affected / at risk) | 0/143 | 0/158
Serious Adverse Events (participants affected / at risk) | 0/143 | 0/158
Other Adverse Events (participants affected / at risk) | 4/143 | 6/158
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | EMC2 (N=143) | Usual Care (N=158)
Medication Side Effects (General disorders) | 4 | 6 — Adverse Events were collected as part of the study battery to identify if the EMC2 intervention was able to monitor and resolve the matter timely should patients experience a side effect.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-09-23): https://cdn.clinicaltrials.gov/large-docs/72/NCT03652272/Prot_SAP_000.pdf